CLINICAL TRIAL: NCT00782899
Title: Prospective Observational Study About Progress of Subjective Well-being Sensation in Schizophrenic Patients
Brief Title: Four Dimensions in Schizophrenia
Acronym: 4D
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Teresa Díez, PhD, Local MC Neuroscience Therapeutic Area Manager, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NES-DUM-2008/2
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2009-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; subjective well-being; depressive symptoms; schizophrenia course
MeSH Terms: conditions — Schizophrenia; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Schizophrenic patients with a acute episode treated in outpatients clinics

SUMMARY:
Observational, non-interventional, longitudinal, prospective,multicenter, open label (No treatment is involved). 4 assessment will be carried out , in months 0, 1, 3 and 6. The primary objective is to asses evolution of subjective well-being and depressive symptoms in schizophrenic patients for six months after an acute episode treated in outpatient psychiatric units. The primary endpoint is: Total score in Subjective Well-being under Neuroleptic treatment (SWN-K) and Calgary Depression Rating Scale (CDRS) scales in assessment after 6 months vs baseline. Secondary objectives include: To evaluate the relationship between subjective well-being and psychopathology, subjective clinical global impression, adverse events and compliance of treatment. Also to compare the clinical global impression of psychiatrist and patient. In addiction to know the clinical, social and demographic factors involve in the subjective well-being and patient clinical global impression.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written inform consent
* Diagnosed of Schizophrenia of Schizoaffective Disorder based on DSM-IV-TR
* With an acute episode or worsening of clinical status. Defined as change in clinical status that need a significant change in therapeutic plan.
* Able to understand and comply with requirements of the study

Exclusion Criteria:

* Mental retardation
* Unstable somatic disease, that is not receiving adequate treatment, based on investigator opinion.
* To have been recruited in a clinical trial in the last 4 weeks
* To have planned the inclusion in a clinical trial during the follow-up of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Schizophrenic patients with a acute episode or worsening of clinical status treated in outpatients clinics. Defined acute episode or worsening as clinical status that need a significant change in the therapeutic plan.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Total score in Subjective Well-being under Neuroleptic treatment (SWN-K) and Calgary Depression Rating Scale (CDRS) scales in assessment after 6 months vs baseline | Months: 0, 1, 3 and 6

SECONDARY OUTCOMES:
Patient Clinical Impression | Months: 0, 1, 3 and 6
Clinical evaluation and social performance | Months: 0, 1, 3 and 6
Adverse events reported by patients | Months: 0, 1, 3 and 6

CONTACTS AND LOCATIONS:
Locations (65):
- Spain (65):
  - Research Site, Vitoria-Gasteiz, Alava
  - Research Site, Almansa, Albacete
  - Research Site, Alcoy, Alicante
  - Research Site, Alicante, Alicante
  - Research Site, Benidorm, Alicante
  - Research Site, El Ejido, Almeria
  - Research Site, Roquetas de Mar, Almeria
  - Research Site, Zafra, Badajoz
  - Research Site, Manacor, Balearic Islands
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Barcelona, Barcelona
  - Research Site, El Hospitalet de Llobregat, Barcelona
  - Research Site, Gavà, Barcelona
  - Research Site, Manresa, Barcelona
  - Research Site, Mataró, Barcelona
  - Research Site, Sabadell, Barcelona
  - Research Site, Sant Feliu de Llobregat, Barcelona
  - Research Site, Santa Coloma de Gramanet, Barcelona
  - Research Site, Terrassa, Barcelona
  - Research Site, Aranda de Duero, Burgos
  - Research Site, Cáceres, Caceres
  - Research Site, Maliaño, Cantabria
  - Research Site, Vinaròs, Castellon
  - Research Site, Donostia / San Sebastian, Guipuzcoa
  - Research Site, Errenteria, Guipuzcoa
  - Research Site, Alcalá la Real, Jaen
  - Research Site, Linares, Jaen
  - Research Site, Logroño, La Rioja
  - Research Site, Banaderos, Las Palmas
  - Research Site, Montforte, Lugo
  - Research Site, Alcalá de Henares, Madrid
  - Research Site, Colmenar Viejo, Madrid
  - Research Site, Fuenlabrada, Madrid
  - Research Site, Getafe, Madrid
  - Research Site, Leganés, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Málaga, Malaga
  - Research Site, Vélez-Málaga, Malaga
  - Research Site, Caravaca de La Cruz, Murcia
  - Research Site, Cartagena, Murcia
  - Research Site, Elizondo, Navarre
  - Research Site, Vigo, Pontevedra
  - Research Site, Arriondas, Principality of Asturias
  - Research Site, Avilés, Principality of Asturias
  - Research Site, Gijón, Principality of Asturias
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Béjar, Salamanca
  - Research Site, Salamanca, Salamanca
  - Research Site, Alcalá de Guadaira, Sevilla
  - Research Site, Écija, Sevilla
  - Research Site, Seville, Sevilla
  - Research Site, Soria, Soria
  - Research Site, El Vendrell, Tarragona
  - Research Site, Reus, Tarragona
  - Research Site, Adeje, Tenerife
  - Research Site, San Cristóbal de La Laguna, Tenerife
  - Research Site, Santa Cruz de Tenerife, Tenerife
  - Research Site, Toledo, Toledo
  - Research Site, Adaia, Valencia
  - Research Site, Catarroja, Valencia
  - Research Site, Mislata, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Valladolid, Valladolid
  - Research Site, Bilbao, Vizcaya
  - Research Site, Zaragoza, Zaragoza